CLINICAL TRIAL: NCT00151138
Title: Cognitive and Cerebrovascular Sequelae of Hypertension
Brief Title: Cognitive/Cerebrovascular Consequences of HTN Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HyperPetII; R01HL057529 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Hypertension
Keywords: cerebral blood flow, positron emission tomography, magnetic resonance imaging, neuropsychology
MeSH Terms: conditions — Hypertension | interventions — Atenolol; Pharmaceutical Preparations; Lisinopril

INTERVENTIONS:
Drug: Atenolol (drug), Lisinopril (drug)

SUMMARY:
Randomized trial of two antihypertensive drugs of known efficacy to investigate whether one has more favorable effects on brain blood flow and cognitive function.

DETAILED DESCRIPTION:
The project examines the neuropsychological status, peripheral blood flow, and structural cortical (magnetic resonance imaging, MRI) and functional cortical blood flow (quantitative positron emission tomography, PET) status of previously unmedicated hypertensives. These individuals are then medicated for one year with one of two effective blood pressure medications. Our hypothesis is that the angiotensin-converting enzyme inhibitor, but not the beta-blocker will normalize cerebral blood flow and possibly, cognitive function. This hypothesis is tested by a repetition of our initial examinations at the completion of one year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be between 35 and 65 years of age, and must have a diastolic BP between 90 and 109 mm Hg, systolic BP between 140 and 179 mm Hg, or both. Eligibility will be based upon readings taken at two screening visits. For resting BP determinations, eating, smoking, drinking and heavy physical activity will be proscribed for 1 hour prior, and drinking caffeinated beverages 2 hours prior. Systolic and diastolic (5th phase) BP will be determined twice separated by 2 minutes using a 2-3 mm Hg/sec deflation rate. Before readings, a 60 s resting pulse will be obtained. Two readings over two such sessions will be averaged. All measurements will be obtained by individuals certified in BP measurement by the Department of Epidemiology of the Graduate School of Public Health.

Potential subjects must have either no prior pharmacologic treatment for hypertension or minimal lifetime exposure. The latter is defined as no more than 6 months of blood pressure medication within the past 5 years. No blood pressure medication taken at all in the 6 months preceding study enrollment. To establish medical eligibility and to screen for secondary causes of hypertension, subjects will provide a medical history and have their standard blood chemistry determined to screen for occult renal failure and primary hyperaldosteronism. All women will be postmenopausal or tested (urine specimen) to ensure the absence of pregnancy. To ensure their ability to complete the behavioral assessments, subjects must have at least an 8th grade education and immigrants must have spoken English as their primary language for at least five years.

Exclusion Criteria. Exclusion criteria will include current use of any cardiovascular or psychotropic medications, or contraindication for use of an ACE inhibitor or beta blocker (e.g., prior adverse reaction or chronic obstructive lung disease, including asthma). Individuals with a resting blood pressure greater than a SBP >180 mmHg and /or a DBP >110 are excluded as are individuals with a prior serious adverse reaction or allergy to beta blockers or angiotensin-converting-enzyme inhibitors. We will exclude individuals with target organ damage (history of myocardial infarction, angioplasty, bypass surgery, congestive heart failure, stroke, or carotid endarterectomy), angina pectoris (determined by Rose questionnaire), a history of insulin-dependent diabetes, or chronic renal insufficiency (serum creatinine > 1.8 mg/dl). Secondary hypertension, based upon known or clinically suspected renal artery stenosis, primary hyperaldosteronism, untreated thyroid disorder, heavy alcohol consumption (24 or more standard drinks per week), consistent use of illegal drugs (for example, crack/cocaine used once or more a month) or pheochromocytoma, will be grounds for exclusion. A standard of no more than 30 g per day (Klatsky, 2003) seems to have some acceptance for the level of alcohol intake that will not chronically alter blood pressure levels. Therefore, no more than a case of beer per week, 21 (5 oz.) glasses of wine, or 21 shots (1.5 oz.) of hard liquor will be acceptable. Exclusion criteria also include neurological disorders (serious head injury, seizures, presenile or alcoholic dementia, Parkinson's disease, or multiple sclerosis). Due to the MRI examination required, individuals not fitting into the bore of the magnet will be excluded. Those with known sensitivity to sulfa-containing antibiotics will be included in the study but will not undergo the acetazolamide portion of the PET scanning sessions: acetazolamide is a sulfonamide analog. Women with child-bearing potential (i.e., pre- or peri-menopausal) will be tested within 48 hours prior to the PET examination to ensure the absence of pregnancy. A urinary pregnancy test (e.g., Sure-Vue Urine hCG) will be administered to confirm the absence of pregnancy.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow in response to working memory task

SECONDARY OUTCOMES:
Neuropsychological function

CONTACTS AND LOCATIONS:
Overall Officials: J. Richard Jennings, PhD, Principal Investigator — University of Pittsburgh, Dept of Psychiatry
Locations (1):
- Dept of Psychiatry, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Jennings JR, Muldoon MF, Ryan C, Price JC, Greer P, Sutton-Tyrrell K, van der Veen FM, Meltzer CC. Reduced cerebral blood flow response and compensation among patients with untreated hypertension. Neurology. 2005 Apr 26;64(8):1358-65. doi: 10.1212/01.WNL.0000158283.28251.3C. PMID 15851723